CLINICAL TRIAL: NCT02488616
Title: An Open-label, Randomized, Two-way, Cross-over Study to Assess the Efficacy of Single-hormone Closed-loop Strategy and Sensor-augmented Pump Therapy in Regulating Glucose Levels for 5 Days in Free-living Outpatient Conditions in Patients With Type 1 Diabetes
Brief Title: Closed-loop Control of Glucose Levels (Artificial Pancreas) for 5 Days in Adults With Type 1 Diabetes
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Medtronic support terminated
Sponsor: Institut de Recherches Cliniques de Montreal (Other)
Responsible Party: Principal Investigator, Rémi Rabasa-Lhoret, Associate Professor of Medicine, Institut de Recherches Cliniques de Montreal
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CLASS-11
Record Dates: First submitted 2015-06-26; First posted 2015-07-02 (Estimated); Last update posted 2018-01-31 (Actual); Status verified 2018-01

CONDITIONS: Type 1 Diabetes
Keywords: Closed-loop system; Artificial pancreas; Type 1 diabetes; Hypoglycemia; Insulin
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Hypoglycemia; Insulin Resistance | interventions — Methods; Insulin Infusion Systems; Continuous Glucose Monitoring; Insulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sensor-augmented pump therapy (Active Comparator): Participants will use sensor-augmented pump therapy with low-glucose suspend to regulate glucose levels. The low-glucose suspend feature available in the MiniMed® Paradigm® Veo™, Medtronic combined with the Enlite sensor® will be used. This feature allows for suspension of insulin delivery at a pre-set sensor glucose value for up to 2 hours.
  Interventions: Other: 5-day intervention with sensor-augmented pump therapy; Device: Insulin pump; Device: Continuous glucose monitoring system; Drug: Insulin
- Single-hormone closed-loop strategy (Active Comparator): Variable subcutaneous insulin infusion will be used to regulate glucose levels. Participant's usual fast-acting insulin analog will be infused using a subcutaneous infusion pump (MiniMed® Paradigm® Veo™, Medtronic). Every 10 minutes, the glucose levels as measured by the sensor (Enlite sensor®, Medtronic) will be transferred automatically to a smartphone, that harbors the algorithm, that will calculate the recommended doses and will send it wirelessly to the infusion pump.
  Interventions: Other: 5-day intervention with single-hormone closed-loop strategy; Device: Insulin pump; Device: Continuous glucose monitoring system; Drug: Insulin

INTERVENTIONS:
Other: 5-day intervention with single-hormone closed-loop strategy — A sensor will be inserted on the day prior to the first day of the intervention by the participants. On the first day of the intervention, participants will be admitted to the clinical research facility anytime between 8:00 am and 11:30 am. Training on connection and disconnection of the system, meal boluses, etc. will be given.
  Competency on the use of study devices will be assessed by a team member. Only participants demonstrating competency on use of study devices will be allowed to continue to the home study phase. Participants will be advised to continue with study intervention at home for the next 5 days.
  Arms: Single-hormone closed-loop strategy
Other: 5-day intervention with sensor-augmented pump therapy — A sensor will be inserted on the day prior to the first day of the intervention by the participants. The participant will also have to install the study insulin pump. Participants will be advised to continue with study intervention at home for the next 5 days.
  Participants will have been previously shown how to use the study insulin pump.
  Arms: Sensor-augmented pump therapy
Device: Insulin pump — MiniMed® Paradigm® Veo™, Medtronic
Device: Continuous glucose monitoring system — Enlite sensor®, Medtronic
Drug: Insulin — Participant's usual fast-acting insulin analog will be used: Lispro (Humalog), Aspart (NovoRapid) or Glulisine (Apidra)

SUMMARY:
Closed-loop strategy is composed of three components: glucose sensor to read glucose levels, insulin pump to infuse insulin and a dosing mathematical algorithm to decide on the required insulin dosages based on the sensor's readings.

The main objective of this project is to compare the efficacy of single-hormone closed-loop strategy and sensor-augmented pump therapy to regulate glucose levels in outpatient settings for 5 consecutive days in adults with type 1 diabetes.

The investigators hypothesized that single-hormone closed-loop strategy will increase the time spent in the target range compared to sensor-augmented pump therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females ≥ 18 years of old.
2. Clinical diagnosis of type 1 diabetes for at least one year.
3. The subject will have been on insulin pump therapy for at least 3 months.
4. HbA1c ≤ 10%.
5. Live in the area of Montreal.

Exclusion Criteria:

1. Clinically significant nephropathy, neuropathy or retinopathy as judged by the investigator.
2. Recent (< 6 months) acute macrovascular event e.g. acute coronary syndrome or cardiac surgery.
3. Warfarin chronic treatment if INR monitoring cannot be evaluated (can increase the risk of bleeding)
4. Pregnancy (ongoing or current attempt to become pregnant).
5. Severe hypoglycemic episode within two weeks of screening.
6. Current use of glucocorticoid medication (except low stable dose and inhaled steroids).
7. Known or suspected allergy to the trial products
8. Other serious medical illness likely to interfere with study participation or with the ability to complete the trial by the judgment of the investigator.
9. Anticipating a significant change in exercise regimen between admissions (i.e. starting or stopping an organized sport).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-03 (Estimated); Primary Completion 2018-11 (Estimated); Study Completion 2018-11 (Estimated)

PRIMARY OUTCOMES:
Percentage of time of glucose levels spent between 3.9 and 10.0 mmol/L | 120 hours

SECONDARY OUTCOMES:
Percentage of time of glucose levels spent between 3.9 and 7.8 mmol/L | 120 hours
Percentage of time of glucose levels spent below 3.9 mmol/L | 120 hours
Percentage of time of glucose levels spent below 3.3 mmol/L | 120 hours
Percentage of time of glucose levels spent below 2.8 mmol/L | 120 hours
Percentage of time of glucose levels spent above 10 mmol/L | 120 hours
Percentage of time of glucose levels spent above 13.9 mmol/L | 120 hours
Percentage of time of glucose levels spent above 16.7 mmol/L | 120 hours
Percentage of time of overnight glucose levels spent below 3.9 mmol/L | 35 hours
Percentage of time of overnight glucose levels spent between 3.9 and 7.8 mmol/L | 35 hours
Percentage of time of overnight glucose levels spent between 3.9 and 10.0 mmol/L | 35 hours
Percentage of time of overnight glucose levels spent below 3.3 mmol/L | 35 hours
Percentage of time of overnight glucose levels spent below 2.8 mmol/L | 35 hours
Percentage of time of overnight glucose levels spent above 10 mmol/L | 35 hours
Percentage of time of overnight glucose levels spent above 13.9 mmol/L | 35 hours
Percentage of time of overnight glucose levels spent above 16.7 mmol/L | 35 hours
Area under the curve of glucose levels below 3.9 mmol/L | 120 hours
Area under the curve of glucose levels below 3.3 mmol/L | 120 hours
Area under the curve of glucose levels below 2.8 mmol/L | 120 hours
Area under the curve of glucose levels above 10 mmol/L | 120 hours
Area under the curve of glucose levels above 13.9 mmol/L | 120 hours
Area under the curve of glucose levels above 16.7 mmol/L | 120 hours
Area under the curve of overnight glucose levels below 3.9 mmol/L | 35 hours
Area under the curve of overnight glucose levels below 3.3 mmol/L | 35 hours
Area under the curve of overnight glucose levels below 2.8 mmol/L | 35 hours
Area under the curve of overnight glucose levels above 10 mmol/L | 35 hours
Area under the curve of overnight glucose levels above 13.9 mmol/L | 35 hours
Area under the curve of overnight glucose levels above 16.7 mmol/L | 35 hours
Mean glucose levels | 120 hours
Standard deviation of glucose levels | 120 hours
Standard deviation of insulin delivery | 120 hours
Coefficient of variance of glucose levels | 120 hours
Coefficient of variance of insulin delivery | 120 hours
Between-day variability in glucose levels | 120 hours
Between-day variability in insulin delivery | 120 hours
Total insulin delivery | 120 hours
Percentage of time of closed-loop operation | 120 hours
Percentage of time of glucose sensor availability | 120 hours
Time between failures | 120 hours
  Total hours of closed-loop operation over number of failures
Number of hypoglycemic events less than 3.1 mmol/L | 120 hours
Number of nights with hypoglycemic events less than 3.1 mmol/L | 35 hours
Number of days with hypoglycemic events less than 3.1 mmol/L | 120 hours

CONTACTS AND LOCATIONS:
Overall Officials: Rémi Rabasa-Lhoret, MD, PhD, Principal Investigator — Institut de recherches cliniques de Montréal
Locations (1):
- Institut de recherches cliniques de Montréal, Montreal, Quebec, Canada